CLINICAL TRIAL: NCT02386579
Title: Characterization of Local and Systemic Bone Markers in Diabetes Patients With Charcot Osteoarthropathy
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Rasmus Bo Jansen, MD, Bispebjerg Hospital
Other Study IDs: H-1-2014-069
Record Dates: First submitted 2015-02-27; First posted 2015-03-12 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Arthropathy, Neurogenic; Diabetes Complications; Diabetes Mellitus
MeSH Terms: conditions — Arthropathy, Neurogenic; Diabetes Complications; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood serum samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diabetics with Charcot foot
  Interventions: Procedure: Blood sample measurements

INTERVENTIONS:
Procedure: Blood sample measurements — Blood samples are drawn in the feet and arms (a/v) before and after cooling the feet with ice water

SUMMARY:
The study is designed to investigate biomarkers related to bone turnover in diabetics with charcot foot. This is done by measuring local blood samples in the feet, and systemically in a vene and an artery. Measurements are done before and after cooling the feet in icewater to lower the bloodflow.

Patients will be compared with healthy diabetic controls.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 1 or 2
* Charcot foot diagnosed with x-ray, scintigraphy or clinical review by a specialist

Exclusion Criteria:

* Osteoporosis
* Anti-osteoporotic treatment
* Lower extremity amputation
* Lower extremity infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diabetes patients with and without acute charcot foot
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-02; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
RANKL | 10 min between measurements

SECONDARY OUTCOMES:
osteocalcin | 10 min between measurements
CTX-I | 10 min between measurements
sRAGE | 10 min between measurements
P1NP | 10 min between measurements